CLINICAL TRIAL: NCT06781294
Title: SIRAKI02 POST-HOC ANALYSIS.
Brief Title: SIRAKI 02 Posthoc Analysis.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: University of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, JOSE LUIS PEREZ FERNANDEZ, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIRAKI02POSTHOC
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass; Acute Kidney Injury; Chronic Kidney Disease(CKD); Kidney Failure, Acute
Keywords: cytokines; heparin; protamine; propofol; vasopressors; insulin; Acute kidney disease; chronic kidney disease; renal recovery; extracorporeal blood purification; hemadsorption; oXiris; cardiopulmonary bypass; cardiac surgery; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION (Active Comparator): Extracorporeal blood purification device connected to cardiopulmonary bypass.
  Interventions: Device: Extracorporeal Cytokine hemadsorption therapy
- CONTROL (No Intervention): Standard of care during cardiopulmonary bypass (includes ultrafiltration with polysulphone if required)

INTERVENTIONS:
Device: Extracorporeal Cytokine hemadsorption therapy — Extracorporeal blood purification with oXiris set connected to cardiopulmonary bypass during all CPB time. Ultrafiltration was permitted.
  Other Names: oXiris; Extracorporeal blood purification device
  Arms: INTERVENTION

SUMMARY:
Our randomized controlled trial with 343 patients requiring non emergent cardiac surgery with a prolonged expected cardiopulmonary bypass (CPB) time (>90 minutes) demonstrated that the use of an extracorporeal blood purification (EBP) device (oXiris) connected to the CPB circuit during all surgery was associated with a decrease in the incidence of CSA-AKI within the first 7 days from surgery (nearly 12% reduction). The study was conducted in two university centres of the Barcelona metropolitan area between 2016 and 2022, randomising 343 patients (1:1) to receive either an EBP device connected to the CPB circuit or a standard strategy with CPB alone.

First of all the rate of acute kidney disease (AKD) and chronic kidney disease (CKD) in the sutdy population has not been reported and we will analyse if there were differences between groups as other studies have suggested with different interventions.

Concerning the intervention safety, no differences were observed in terms of intraoperative blood products (red blood cells, plasma and platelets) requirements between both groups. In order to improve knowledge about the safety of the technique it is very important to ensure that antibiotics levels in plasma during the time the adsorption device is connected to CPB, are not being modified by the intervention. Antibiotic prophylaxis during cardiac surgery is one of the cornerstones and has proved to effectively reduce perioperative infection especially concerning valve replacement procedures. In this sense, our two centres use the same strategy with cephalosporins (Cefazolin in Germans Trias Hospital and Cefuroxime in Bellvitge Hospital) with an early administration at the operating room (OR) before connecting patient to CPB and a late dose after removing CPB (3 hours after the first dose). We know from previous reports that the use of antibiotics during CRRT with oXiris is safe and normally does not require dose adjustments although no reports have been made of its use connected to CPB and antibiotics dosing.

Completing the safety issues, heparin and protamine doses during surgery have been registered in the patient's electronic history and should be checked and transferred to a database that allows to adequately analyse potential differences between groups. Other studies performed in cardiac surgery with adsorption devices have reported safety issues with platelets consumption and heparin requirements during surgery. In our protocol, heparin was administered prior to CPB initiation either based on the patient's weight or using hemostasis management system (HMS) plus technology in order to minimise overdosing. Heparin was administered during all CPB time in order to maintain activated clotting time (ACT) over 500 seconds and based on HMS plus technology. Protamine for heparin reversal at CPB withdrawal was administered using both methods too. Protamine administration can be associated with hypotensive episodes.

In our study, the decrease in CSA-AKI within the first 7 days from surgery achieved with the use of EBP connected to the CPB was more significant in CKD, DM, Low LVEF, Hypertension and non-obese patients. Whether this effect can be partially explained by the mild cytokines concentration differences observed in IL-8 and TNF-a at T1 (after removing clamp from surgery) and T2 (at ICU admission) has still not been evaluated. This reduction of inflammatory response syndrome (SIRS) during CPB time that could be related with the use of adsorption devices, should be also translated into a decrease of catecholamines and probably insulin requirements during surgery.

A noteworthy point to consider is that although the use of propofol has been extended in cardiac surgery, little is known about the potential antiinflammatory effect it may have in patients. It is important to identify those patients who received propofol to control this potential bias in terms of antiinflammatory effect. Besides this objective it is also very important to ensure that no adsorption of propofol took place with the use of EBP, as previous studies have reported higher requirements of sedation drugs with the use of CRRT or other devices with adsorption properties.

Finally, nearly 25% of the patients in the EBP group received ultrafiltration with doses that vary from 200 mL up to 3000 mL. We know from previous trials that ultrafiltration is clearly related with the removal of middle weight molecules which is presumably beneficial for patients with SIRS but that in specific scenarios this effect could be even detrimental for some patients. Whether the ultrafiltration performed in our study may have an effect in antibiotics, heparin, protamine, catecholamines, insulin or even propofol should be elucidated in order to settle the idoneous modality in which EBP should be performed when connected to CPB during cardiac surgery.

All these outcomes will be assessed controled by gender and age.

DETAILED DESCRIPTION:
The study was conducted in two university centres of the Barcelona metropolitan area between 2016 and 2022 randomising 343 patients (1:1) to receive either an intervention strategy with EBP connected to the CPB circuit (169 patients) or a standard strategy with CPB alone (174 patients).

Cefuroxime was employed as antibiotic prophylaxis in 223 patients and Cefazolin was employed as antibiotic prophylaxis in the other 120 patients. These variations were due to the different hospital protocols for cardiac surgery antibiotic prophylaxis.

In 205 patients (111 in the control group and 94 in the EBP group), we recollected blood samples that were centrifuged, aliquoted and stored at -70º Celsius. 119 patients received Cefazolin protocol prophylaxis and 86 patients received Cefuroxime protocol prophylaxis. The samples from these patients were obtained at the beginning of the surgical intervention (T0), at the clamp withdrawal (T1), at the ICU admission (T2) and 24 hours after (T3). To evaluate the primary endpoint, antibiotic mass concentrations in plasma samples from T1 checkpoint will be measured using a previously validated ultra-high-performance liquid chromatography-tandem mass spectrometry method (Rigo-Bonnin R, Ribera A, Arbiol-Roca A, et al. Development and validation of a measurement procedure based on ultra-high performance liquid chromatography-tandem mass spectrometry for simultaneous measurement of β-lactam antibiotic concentration in human plasma. Clin Chim Acta. 2017;468:215-24).

In all patients (343 patients, 174 in the control group and 169 in the EBP group), we have planned to complete collecting all the hemodynamic and respiratory data in the operating room (OR) besides all the drugs administered in the OR (antibiotics, heparin, protamine, norepinephrine, insulin, and propofol). Laboratory parameters during surgery will be obtained from the medical records. Specific CPB parameters and ultrafiltration data when performed will also be collected. Kidney function parameters (creatinine and other biomarkers) will be registered up to 90 days after cardiac surgery and CKD incidence will be monitored up to 1 year after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non emergent cardiac surgery requiring cardiopulmonary bypass with expected CPB time over 90 minutes (double valve replacement or valve replacement plus CABG).
* Written informed consent from patient or legal surrogates.

Exclusion Criteria:

* Transplant receptor.
* Advanced Chronic Kidney Disease (CKD 4 or 5).
* Renal replacement therapy in the last 90 days.
* Documented intolerance to study device.
* Inclusion in other ongoing study within the last 30 days.
* Pregnancy.
* Immunosuppressive treatment or steroids (prednisone > 0.5 mg/kg/day or equivalent).
* Autoimmune disorder.
* Coexisting illness with a high probability of death (inferior to 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Cytokines differences in subgroups | 24 hours
  Cytokine differences (IL-2, IL-6, IL-8, IL-10, TNF-a, and INF-y) between intervention and standard care in subgroups (CKD, Low LVEF, DM, Hypertension and non-obese population). Determination of cytokines was done at baseline (T0), end of CPB (T1), ICU admission (T2), and 24 hours after surgery (T3). Variations of these cytokines levels (especially during CPB T1-T0) will be analysed in subgroups where the intervention with the EBP device seemed to be more effective.

SECONDARY OUTCOMES:
Intraoperatory antibiotic concentrations. | During surgery
  Cefuroxime and Cefazolin antibiotic concetrations will be determined at T1 (end of cardiopulmonary bypass) to evaluate differences between both groups.
Heparin administration | During surgery
  Differences in heparin administered (total milligrams) during all cardiopulmonary bypass time.
Protamine administration. | During surgery
  Protamine administration differences (total milligrams) between groups during surgery.
Insulin subcutaneous administration. | During surgery
  Insulin subcutaneous administration (total international units) differences between groups during cardiac surgery.
Vasopressor administration (Norepinephrine). | During surgery
  Vasopressor administration differences between groups during cardiac surgery. Norepinephrine total micrograms administered will be registered during all surgery.
Propofol administration. | During surgery
  Propofol administration differences (total milligrams) between groups during cardiopulmonary bypass time.
Acute Kidney Disease rate | 90 days
  Rate of acute kidney disease (AKD) and differences between groups. AKD is defined as the persistence of acute kidney injury (AKI) beyond day 7 and up to 90 days after AKI. Creatinines will be registered in all patients up to day 90.
Chronic Kidney Disease (CKD) rate. | One year
  Rate of Chronic kidney disease (CKD) and differences between groups. CKD is defined as a glomerular filtration rate (GFR) under 60 mL/min more than 90 days after AKI. GFR will be registered in all patients up to one year after cardiac surgery.
PenKid and BioADM determinations. | 24 hours
  PenKid and BioADM concentrations will be measured at T1 (end of cardiopulmonary bypass time) to determine the usefulness of these two biomarkers to detect AKI, AKD and CKD.
Urinary CCL-14 evaluation. | During surgery
  CCL-14 urinary evaluation will be performed at T1.
Adsorption circuit blood flow | During surgery.
  Adsorption circiut blood flow rates and their correlation with CSA-AKI will be analysed in order to identify optimal blood flow rates.
Ultrafiltration rates | During surgery.
  Ultrafiltration rates in those patients ultrafiltrated will be analysed in oder to evaluate their impact in primary and secondary outcomes such as cytokines or antibiotic concentrations.
EBP time and Clamp time. | During surgery.
  Relationship between time on EBP and time with clamp will be analysed in those patients assigned to the EBP group. Preliminary analysis revealed that clamp time seem to be protective in terms of CSA-AKI incidence in the EBP group and this could be related to an early withdrawal of the EBP circuit after clamp removal. If this effect is demonstrated we should suggest to maintain the EBP circiut until the end of CPB.
Delirium during ICU stay | 7 days
  Presence of delirium during the first 7 days after cardiac surgery defined by CAM-ICU criteria. Criteria will be evaluated every day besides administration of haloperidol (mg/day) and / or dexmedetomidine (mg/day).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Fernandez X, Ulsamer A, Camara-Rosell M, Sbraga F, Boza-Hernandez E, Moret-Ruiz E, Plata-Menchaca E, Santiago-Bautista D, Boronat-Garcia P, Gumucio-Sanguino V, Penafiel-Munoz J, Camacho-Perez M, Betbese-Roig A, Forni L, Campos-Gomez A, Sabater-Riera J; SIRAKI02 Study Group. Extracorporeal Blood Purification and Acute Kidney Injury in Cardiac Surgery: The SIRAKI02 Randomized Clinical Trial. JAMA. 2024 Nov 5;332(17):1446-1454. doi: 10.1001/jama.2024.20630. PMID 39382234